CLINICAL TRIAL: NCT06261580
Title: Procedure to Define a Normal Reference Range Using the TEG® 6s Diagnostic System With the Heparin Neutralization Cartridge in Healthy Volunteers
Brief Title: Normal Reference Range Study With the TEG6s Heparin Neutralization Cartridge in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Haemonetics Corporation (Industry)
Collaborators: Machaon Diagnostics (Industry); ClinStatDevice (Unknown)
Responsible Party: Sponsor
Other Study IDs: TP-CLN-100502
Record Dates: First submitted 2023-03-31; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Adult volunteers (18 years of age and older) who self-identify as being in general good health were recruited at 3 US centers. Whole Blood Samples and frozen plasma were collected for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Healthy Volunteers: Adult volunteers (18 years of age and older) who self-identify as being in general good health.
  Interventions: Diagnostic Test: TEG 6s Citrated K, KH, RTH, and FFH Cartridge; Diagnostic Test: Clauss Fibrinogen

INTERVENTIONS:
Diagnostic Test: TEG 6s Citrated K, KH, RTH, and FFH Cartridge — The TEG® 6s uses the Global Hemostasis with Heparin Neutralization (HN) Cartridge to test the hemostasis properties of citrated blood samples using four different assays/reagents simultaneously, one in each of the four cartridge channels.
Diagnostic Test: Clauss Fibrinogen — Fibrinogen, also known as Factor I, is a plasma protein that can be transformed by thrombin into a fibrin gel ("the clot"). Fibrinogen is synthesized in the liver and circulates in the plasma as a disulfide-bonded dimer of 3 subunit chains. The biological half-life of plasma fibrinogen is 3 to 5 days.

SUMMARY:
This trial holds minimal risk to the trial volunteers and consists of obtaining whole blood via venipuncture to perform coagulation parameter measurements to define a Normal Reference Range.

Written consent to participate in the study will be obtained prior to volunteer screening per site procedures.

ELIGIBILITY:
Inclusion Criteria:

• Adult volunteers (18 years of age and older) who self-identify as being in general good health.

Exclusion Criteria:

* Volunteers with any acute illness or uncontrolled chronic disease
* Volunteers with any type of cancer
* Volunteers with diabetes
* Volunteers with renal disease
* Volunteers with liver disease
* Volunteers with morbid obesity
* Volunteers with autoimmune or inflammatory diseases
* Volunteers with known coagulation and/or bleeding disorders (e.g., hemophilia, Von Willebrand's disease)
* Volunteers currently abusing alcohol (defined as more than 3 drinks for women and more than 4 drinks for men on any given day, or 7 drinks for women and 14 drinks for men throughout the week) or taking illicit drugs
* Volunteers with hereditary fibrinolytic bleeding disorders
* Volunteers with altered coagulation due to the presence of direct oral anticoagulants (e.g., apixaban, rivaroxaban, dabigatran) in the blood
* Volunteers on any fibrinolytic activators (e.g., Streptokinase, t-PA, Reteplase, Tenecteplase, Urokinase, APSAC, Staphylokinase)
* Volunteers who have had recent surgery (within the last four weeks)
* Volunteers with any injuries leading to substantial bleeding or bruising (within the last two weeks prior to blood donation)
* Volunteers with bruising, wounds, or scarring around the selected venipuncture site
* Volunteers deemed unfit for participation in the trial by the principal investigator
* Volunteers participating in another clinical trial that would not be scientifically or medically compatible with this trial
* Volunteers who have been on P2Y12 inhibitors within the last 30 days
* Volunteers receiving treatment with low molecular weight heparin (e.g., enoxaparin)
* Volunteers with altered coagulation due to the presence of drugs known to affect the coagulation status in the blood (see Table 1)
* Volunteers who have participated in this trial previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
CK-MA TEG Parameter | Outcome measure from the single blood draw was assessed within 2 hours of blood draw. Unit of measurement was mm.
  Citrated Kaolin Maximum Amplitude Thromboelastographic Result
CK-R TEG Parameter | Outcome measure from the single blood draw was assessed within 2 hours of blood draw. Unit of measurement was minutes.
  Citrated Kaolin Reaction Time Thromboelastographic Result
CKH-MA TEG Parameter | Outcome measure from the single blood draw was assessed within 2 hours of blood draw. Unit of measurement was mm.
  Citrated Kaolin with Heparinase Maximum Amplitude Thromboelastographic Result
CKH-R TEG Parameter | Outcome measure from the single blood draw was assessed within 2 hours of blood draw. Unit of measurement was minutes.
  Citrated Kaolin with Heparinase Reaction Time Thromboelastographic Result
CKH-LY30 TEG Parameter | Outcome measure from the single blood draw was assessed within 2 hours of blood draw. Unit of measurement was percentage.
  Citrated Kaolin with Heparinase Lysis Thromboelastographic Result
CRTH-MA TEG Parameter | Outcome measure from the single blood draw was assessed within 2 hours of blood draw. Unit of measurement was mm.
  Citrated Rapid TEG with Heparinase Maximum Amplitude Thromboelastographic Result
CFFH-MA TEG Parameter | Outcome measure from the single blood draw was assessed within 2 hours of blood draw. Unit of measurement was mm.
  Citrated Rapid TEG with Heparinase Maximum Amplitude Thromboelastographic Result

CONTACTS AND LOCATIONS:
Overall Officials: Yamini Bynagari, PhD, Principal Investigator — Machaon Diagnostics
Locations (3):
- United States (3):
  - Machaon Diagnostics, Oakland, California
  - Cardiovascular Research Institute - Loyola University Chicago Health Sciences, Maywood, Illinois
  - Louisiana Coagulation / Machaon Division, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No